CLINICAL TRIAL: NCT03690765
Title: Observational Open-Label Multicenter Study of Real Clinical Practice to Evaluate the Effects of Hormonal Therapy With Oral Dydrogesterone for Treatment of Confirmed Endometriosis (ORCHIDEA)
Brief Title: Study of Real Clinical Practice to Evaluate the Effects of Oral Dydrogesterone for Treatment of Confirmed Endometriosis
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: DYDR5004
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2019-06

CONDITIONS: Endometriosis
Keywords: endometriosis; dydrogesterone; Duphaston®; progestogens; pelvic pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Dydrogesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometriosis/Dydrogesterone: Females aged 18 to 45 years, suffering external genital endometriosis confirmed by laparoscopy, for whom were prescribed treatment with Duphaston®
  Interventions: Drug: Duphaston® (Dydrogesterone)

INTERVENTIONS:
Drug: Duphaston® (Dydrogesterone) — No intervention. Duphaston® is prescribed according local labelling for treatment of endometriosis 10 mg 2-3 times a day from the 5th to the 25th day of the menstrual period cycle. Description of routine practice only.
Drug: Duphaston® (Dydrogesterone) — No intervention. Duphaston® is prescribed according local labelling for treatment of endometriosis 10 mg 2-3 times a day continuously. Description of routine practice only.

SUMMARY:
A non-interventional, observational program to assess the effects of dydrogesterone (Duphaston®) 6-months-administration in patients with confirmed endometriosis in a post-marketing setting in the Russian Federation

DETAILED DESCRIPTION:
A non-interventional, observational program to assess the effects of oral dydrogesterone therapy in a post-marketing setting whether the effects are related to the regimen of dydrogesterone therapy. In this observational program, assuming that dydrogesterone plays a role in the treatment of endometriosis without suppression of ovulation, the goal is to observe the possible implications of such treatment in terms of treatment regimen and response pattern. In the study will be described effects of Duphaston® 6-months-administration in patients with confirmed endometriosis by assessing pain relief, quality of life, need of self-medication with analgesics, etc.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥ 18 years and ≤ 45 years.
* Complaints on chronic pelvic pain with or without dysmenorrhea assessed by 11-items NRS.
* External genital endometriosis confirmed by laparoscopy.
* Existing pelvic (vaginal) ultrasound data not earlier than 2 months before inclusion in the study.
* Prescribed treatment with Duphaston® according local labelling for treatment of endometriosis 10 mg 2-3 times a day from the 5th to the 25th day of the menstrual period cycle or continuously.
* No hormonal treatment in 2 cycles before enrollment.
* Signed Patient Authorization for Use/Disclosure of Data.

Exclusion Criteria:

* Any co-existing disease(s) needing chronic drug therapy (e.g. Crohn's disease, diabetes etc); Severe concomitant medical illness.
* Severe other genital pathology excluding endometriosis (e.g. Multiple/severe myoma; adenomyosis, inflammatory diseases, etc.).
* Routine consumption of analgesics other than for the pain of endometriosis.
* Patients receiving hormonal contraceptives in last 2 cycles (including intrauterine devices, contraceptive patches, contraceptive rings, oral contraceptives etc.).
* Ongoing pregnancy.
* Menopause or premature ovarian failure.
* Contraindications to dydrogesterone treatment listed in the locally approved label (Instructions for the medical use of Duphaston®).
* Any other condition that precludes use of dydrogesterone in a particular patient, in accordance with the precautions and special warnings listed in the locally approved label (Instructions for the medical use of Duphaston®).
* Abnormal results of pap smear test.
* Other conditions that made the patients participation impossible (based on the investigator decision).
* Fertility treatments using assisted reproductive technology.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Females aged 18 to 45 years, suffering external genital endometriosis confirmed by laparoscopy, for whom were prescribed treatment with Duphaston®
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Change in chronic pelvic pain intensity | 6 months
  The changes in chronic pelvic pain intensity assessed by 11-items Numerous Rating Scale (NRS) at the end of observation (Visit 3) versus Baseline (Visit 1) in the prolonged cyclic regime and the continuous regime of Duphaston in patients with endometriosis. The 11-items Numerous Rating Scale (NRS) contains the range from 0 to 10, where 0 represents 'no pain' and 10 represents 'the worst pain'. Patients are asked to point the average pain intensity throughout the last month. The negative change corresponds to better result.

SECONDARY OUTCOMES:
Change in Quality of Life | 3 months, 6 months
  Changes in Quality of Life assessed by Short Form-20 (SF-20) at the end of observation (Visit3) versus Baseline (Visit1) in patients with endometriosis. The Short Form-20 (Copyright © the RAND Corporation) consists of 20 questions grouped into two parameters: psychological and physical components of health. The indicators of each scale are compiled in such a way that the higher the value of the indicator (from 0 to 100), the better the score on the chosen parameter.
Change in chronic pelvic pain intensity | 3 months, 6 months
  Change in Patient-reported severity of chronic pelvic pain assessed by 11-items NRS after 3-months treatment (Visit2) and after 6-months treatment (Visit3) versus Baseline (Visit1) in patients with endometriosis
Cycles' duration | 6 months
  Description of the cycles' duration during 6-months treatment by Duphaston® in patients with endometriosis
Change in dysmenorrhea | 3 months, 6 months
  Description of the changes in dysmenorrhea assessed by 11-items NRS after 3-months treatment (Visit2) and after 6-months treatment (Visit3) versus Baseline (Visit1) in patients with endometriosis. The 11-items Numerous Rating Scale (NRS) contains the range from 0 to 10, where 0 represents 'No symptoms' and 10 represents 'the Worst trouble'. Patients are asked to point the average intensity of dysmenorrhea symptoms (cyclic pelvic pain, mood disorders, gastro-intestinal symptoms etc.) during the last menses period. The negative change corresponds to better result.
Analgesics using | 6 months
  A number of days per each cycle (1-6) when analgesics were self-administered
Sexual wellbeing | 6 months
  Description of the change in sexual wellbeing assessed by A Quality Assessment of Patient-Reported Outcome Measures for Sexual Wellbeing (5-points Likert scale) at the end of observation (Visit3) versus Baseline (Visit1). A Quality Assessment of Patient-Reported Outcome Measures for Sexual Wellbeing by 5-points Likert scale proposes patients to rate themselves on a 5-point scale as being 'very satisfied, satisfied, ordinarily, rather not satisfied, not satisfied'. The number (and proportion) of patients in each category will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey V Kozachenko, Prof, Study Chair — Kulakov National Medical Research Center of Obstetrics, Gynecology and Perinatology
Locations (20):
- Russia (20):
  - South Ural State Medical University, Department of Obstetrics and Gynecology, Chelyabinsk
  - Engels Perinatal Center, Engel's
  - City Hospital №11, Kazan'
  - Kemerovo State Medical University, Reshetov Kemerovo Regional Perinatal Center, Kemerovo
  - Kuban State Medical University. Regional Clinical Hospital №2, Krasnodar
  - Voyno-Yasenetsky Krasnoyarsk State Medical University, Krasnoyarsk Regional Clinical Center for the Protection of Motherhood and Childhood, Krasnoyarsk
  - Voyno-Yasenetsky Krasnoyarsk State Medical University, Professorial clinic, Krasnoyarsk
  - RZD Central Clinical Hospital № 6, Moscow
  - Kulakov National Medical Research Center of Obstetrics, Gynecology and Perinatology, Moscow
  - Clinical Center for Family Health and Reproduction of the Novosibirsk Region, Novosibirsk
  - Rostov State Medical University, Research institute of obstetrics and pediatrics, Rostov-on-Don
  - Pavlov First St. Petersburg State Medical University, Saint Petersburg
  - Ott Research Institute of Obstetrics, Gynecology and Reproductology, Saint Petersburg
  - Stavropol State Medical University, Stavropol
  - State Hospital Perinatal Center, Tyumen
  - Bashkir State Medical University, Ufa
  - Semashko Nizhny Novgorod Regional Clinical Hospital, Veliky Novgorod
  - Clinic "New Medical Technologies", Voronezh
  - Voronezh Regional Clinical Hospital №1, Voronezh Regional Perinatal Center, Voronezh
  - FOTEK Medical Holding LLC, Women's Clinic, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sukhikh GT, Adamyan LV, Dubrovina SO, Baranov II, Bezhenar VF, Kozachenko AV, Radzinsky VE, Orazov MR, Yarmolinskaya MI, Olofsson JI. Prolonged cyclical and continuous regimens of dydrogesterone are effective for reducing chronic pelvic pain in women with endometriosis: results of the ORCHIDEA study. Fertil Steril. 2021 Dec;116(6):1568-1577. doi: 10.1016/j.fertnstert.2021.07.1194. Epub 2021 Aug 28. PMID 34465452